CLINICAL TRIAL: NCT04081220
Title: An Investigator Initiated Phase 2 Trial of the LSD1 Inhibitor IMG-7289 in Essential Thrombocythemia (CTMS# 19-0078)
Brief Title: Hematology, IMG-7289, LSD1 (Lysine-Specific Demethylase 1) Inhibitor, Essential Thrombocythemia (ET), Ph 2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 19-0078; HSC20190791H (Other: UT Health Science Center San Antonio IRB)
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Thrombocythemia, Essential
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — bomedemstat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMG-7289 (Experimental)
  Interventions: Drug: IMG-7289

INTERVENTIONS:
Drug: IMG-7289 — Single starting dose with individualized dose titrations throughout
  Other Names: LSD1 inhibitor

SUMMARY:
This is a single-center, open-label investigator-initiated trial evaluating the effects of IMG-7289 administered orally once daily in patients with essential thrombocythemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of Essential Thrombocythemia per World Health Organization (WHO) diagnostic criteria for myeloproliferative neoplasms (Arber et al., 2016).
* 3. Patients who are intolerant or resistant to hydroxyurea per ELN (European Leukemia Net) criteria, or in the Investigator's judgment are not candidates for available approved therapy. The ELN definitions of resistance/intolerance to HU (hydroxyurea) requires the fulfillment of at least one of the following criteria:

  * Platelet count greater than 600 × 109/L after 3 months of at least 2 g/day of HU (2.5 g/day in patients with a body weight over 80 kg);
  * Platelet count greater than 400 × 109/L and leukocytes less than 2.5 × 109/L or hemoglobin (Hb) less than 100 g/L at any dose of HU;
  * Presence of leg ulcers or other unacceptable mucocutaneous manifestations at any dose of HU;
  * HU-related fever.
* Requires treatment in order to lower platelet counts based on the Clinically Relevant IPSET (International Prognostic Score for Thrombosis in Essential Thrombocythemia) -Thrombosis Guidelines.
* Platelet count >450 x 109/L pre-dose Day 1.
* Peripheral blast count <10% pre-dose Day 1.
* ANC (absolute neutrophil count) ≥0.5 x 109/L pre-dose Day 1.
* Fibrosis Score ≤ grade 2, as per a slightly modified version (Arber et al., 2016) of the European Consensus Criteria for Grading Myelofibrosis, (Thiele et al., 2005).
* Life expectancy > 36 weeks.
* Able to swallow capsules.
* Amenable to spleen size determination, bone marrow evaluations, and peripheral blood sampling during the study.
* Must have discontinued ET therapy at least 2 weeks (4 weeks for interferon) prior to study drug initiation.
* Agrees to use an approved method of contraception from Screening until 28 days after last administration of the study drug. Acceptable methods of birth control include: birth control pills, depo-progesterone injections, a vaginal hormonal contraceptive ring, a barrier contraceptive such as a condom with spermicide cream or gel, diaphragms or cervical cap with spermicide cream or gel, or an intrauterine device (IUD).
* If male, agrees not to donate sperm or father a child for at least one month after the last dose of the study medication.

Exclusion Criteria:

* Greater than 3 separate transfusion episodes over the last 6 months and/or any transfusion over the last 4 weeks.
* Eastern Cooperative Oncology Group (ECOG) questionnaire score of 3 or greater.
* Currently pregnant or planning on being pregnant in the following 6 months or currently breastfeeding.
* Currently residing outside the United States.
* History of splenectomy.
* Unresolved treatment related toxicities from prior therapies (unless resolved to ≤ Grade 1).
* Uncontrolled active infection.
* Known positive for HIV or infectious hepatitis, type A, B or C.
* Current use of monoamine oxidase A and B inhibitors (MAOIs).
* Evidence at the time of screening of increased risk of bleeding, including any of the following:

  1. Activated partial thromboplastin time (aPTT) > 1.3 x the upper limit of normal
  2. International normalized ratio (INR) >1.3 x the local upper limit of normal
  3. Known Acquired Von Willebrand's disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2026-12-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zohra Nooruddin, MD, Principal Investigator — Mays Cancer Center
Locations (1):
- Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMG-7289
Started | 9
Completed | 5
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Participants enrolled and assigned to treatment
Arm/Group | IMG-7289
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Achieve Complete Hematologic Remission at Week 24 Using ELN Response Criteria for ET (Barosi et al., 2013)
Description: ELN criteria
Time Frame: 24 weeks
Population: Only 4 of the 5 completers were evaluable.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMG-7289
Number analyzed (Participants) | 4
Percentage of Participants | 0

2. Secondary Outcome: Additional Therapy Period (ATP) Overall Symptom Burden
Description: Symptom Forms will be completed by participants each week of participation in the study- even on weeks with no study visit. Symptom Form are completed at around the same time on each of the following days: Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50, Day 57, Day 64, Day 71, Day 78, Day 85, Day 92, Day 99, Day 106, Day 113, Day 120, Day 127, Day 134, Day 141, Day 148, Day 155, Day 162 and Day 169.
Time Frame: 24 weeks to 48 weeks (may repeat)
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: AEs are assessed through regular investigator assessments and laboratory testing.
Arm/Group | IMG-7289
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMG-7289 (N=9)
Nausea (Gastrointestinal disorders) | 1 (1) — Nausea, hyponatremia and generalized muscle weakness
Hyponatremia (Renal and urinary disorders) | 1 (1) — Grade 3 Hyponatremia
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMG-7289 (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 5 (9)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (9)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fatigue (General disorders) | 4 (10)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Malaise (General disorders) | 3 (4)
Memory impairment (Nervous system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (13)
Neutrophil count decreased (Investigations) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Seizure (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
COVID 19 (Infections and infestations) | 1 (1)
Fever (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Uterine Cramp (Reproductive system and breast disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Bursitis Left Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Abscess cheek (Infections and infestations) | 1 (1)
Low Back Spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased red blood cells (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04081220/Prot_SAP_000.pdf